CLINICAL TRIAL: NCT01361698
Title: Illness Management and Recovery (IMR) in Danish Community Mental Health Centres: Protocol of a Randomized, Assessor-blinded Multi-centre Clinical Trial of a Recovery-oriented Program for People With Schizophrenia or Bipolar Disorder
Brief Title: Illness Management and Recovery (IMR) in Danish Community Mental Health Centres
Acronym: IMR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amager Hospital (Other)
Collaborators: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other); The Danish Health Fund (Unknown)
Responsible Party: Principal Investigator, Lene Falgaard Eplov, Head of Research, Associate professor, Amager Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2010B114; IMR-DP-228-CT-59 (Registry Identifier: Copenhagen Trial Unit)
Record Dates: First submitted 2011-05-25; First posted 2011-05-27 (Estimated); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Schizophrenia; Bipolar Disorder
Keywords: recovery; illness management; rehabilitation; mental illness; psychosocial intervention; Clinical recovery (increase in functioning, decrease in symptoms); Personal recovery (Hope, optimism, living a fulfilling life)
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Mental Disorders | interventions — Salvage Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IMR program (Experimental): The program is organised into 11 curriculum topic areas: recovery strategies, practical facts about mental illness, the stress-vulnerability model, building social support, using medication effectively, drug and alcohol use, reducing relapses, healthy lifestyle, coping with stress, coping with problems and symptoms, and getting your needs met in the mental health system. In this Danish trial IMR will be implemented in group format with 10 patients assigned to each group and two IMR facilitators, and the IMR program will require nine months of weekly sessions to complete.
  Interventions: Behavioral: Illness Management and Recovery (IMR)
- Treatment as usual (No Intervention): Patients randomised to the control group will get 'treatment as usual' only. This means individual adapted interdisciplinary treatment including medication, individual support, occupational therapy, psycho-education and group therapy.

INTERVENTIONS:
Behavioral: Illness Management and Recovery (IMR) — In this Danish trial IMR will be implemented in group format with 10 patients assigned to each group and two IMR facilitators, and the IMR program will require nine months of weekly sessions to complete.
  Arms: IMR program

SUMMARY:
The aim of this trial is to evaluate the effectiveness of the Illness Management and Recovery program for people diagnosed with schizophrenia or bipolar disorder in according to their level of functioning.

DETAILED DESCRIPTION:
Background: Illness Management and Recovery (IMR) is a curriculum-based psychosocial intervention designed as structured program with a recovery-oriented approach. The aim of IMR is to rehabilitate people with severe mental illnesses by helping them acquire knowledge and skills in managing their illness and achieve personal recovery goals. Previous randomised clinical trials indicate that IMR can be implemented with a good effect and a high fidelity though further trials are crucial to demonstrate the potential effectiveness of IMR.

Methods/Design: The trial design is a randomised, assessor-blinded, multi-centre, clinical trial of the IMR program compared with treatment as usual for 200 participants diagnosed with schizophrenia or bipolar disorder under the care of two community mental health centres in the Capital Region of Denmark. The primary outcome is level of functioning at the end of treatment and at follow-up 21 months after baseline. The secondary outcomes are disease symptoms; use of alcohol/drugs; individual meaning of recovery; hope; hospital admissions and out-patient psychiatric treatment at the end of treatment and at follow-up 21 months after baseline.

ELIGIBILITY:
Inclusion Criteria:

* adults (age 18+)
* both sexes
* associated with one of the two participating community mental health centres
* diagnosed following the ICD-10 criteria of schizophrenia or bipolar disorder
* able to speak and understand Danish
* giving informed consent verbally and in writing

Exclusion Criteria:

* have a guardian or a forensic psychiatric arrangement
* comorbidity with the ICD-10 criteria of the diagnoses of dementia or mental retardation
* a large-scale substance abuse - if later on the abuse is under control inclusion in the trial will be possible
* a current home of supported housing - since the treatment as usual given to this group of patients is significant different from patients living independently
* a current involvement in a psycho-educational course - patients are eligible for participation in the trial after the psycho-educational course has ended if they meet the inclusion criteria at this point
* not given informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2011-02; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Global Assessment of Function | 9 months and 21 months

SECONDARY OUTCOMES:
PANSS | 9 and 21 months follow-up
  Positive and Negative Syndrome Scale
IMR Scale | 9 and 21 months follow-up
Personal and Social Performance | 9 and 21 months
Hamilton Rating Scale for Depression | 9 & 21 months
Young Mania Rating Scale | 9 & 21 months
Mental Health Recovery Measure | 9 and 21 months
The Adult State Hope Scale | 9 and 21 months

CONTACTS AND LOCATIONS:
Locations (1):
- Community Mental Health Center Ballerup and Community Mental Health Center Frederiksberg, Ballerup and Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mueser KT, Corrigan PW, Hilton DW, Tanzman B, Schaub A, Gingerich S, Essock SM, Tarrier N, Morey B, Vogel-Scibilia S, Herz MI. Illness management and recovery: a review of the research. Psychiatr Serv. 2002 Oct;53(10):1272-84. doi: 10.1176/appi.ps.53.10.1272. PMID 12364675
- [Background] Mueser KT, Meyer PS, Penn DL, Clancy R, Clancy DM, Salyers MP. The Illness Management and Recovery program: rationale, development, and preliminary findings. Schizophr Bull. 2006 Oct;32 Suppl 1(Suppl 1):S32-43. doi: 10.1093/schbul/sbl022. Epub 2006 Aug 9. PMID 16899534
- [Derived] Jensen SB, Dalum HS, Korsbek L, Hjorthoj C, Mikkelsen JH, Thomsen K, Kistrup K, Olander M, Lindschou J, Mueser KT, Nordentoft M, Eplov LF. Illness management and recovery: one-year follow-up of a randomized controlled trial in Danish community mental health centers: long-term effects on clinical and personal recovery. BMC Psychiatry. 2019 Feb 11;19(1):65. doi: 10.1186/s12888-019-2048-0. PMID 30744590
- [Derived] Dalum HS, Korsbek L, Mikkelsen JH, Thomsen K, Kistrup K, Olander M, Hansen JL, Nordentoft M, Eplov LF. Illness management and recovery (IMR) in Danish community mental health centres. Trials. 2011 Aug 17;12:195. doi: 10.1186/1745-6215-12-195. PMID 21849024
- See also: Illness management and recovery (IMR) in Danish community mental health centres (Study protocol) — http://www.trialsjournal.com/content/12/1/195